CLINICAL TRIAL: NCT02352168
Title: To Evaluate Airway Inflammation in Children With Allergic Rhinitis and To Examine the Effects of Nasal Corticosteroids Therapy on Lower Airway Inflammation of Rhinitis.
Brief Title: Airway Inflammation in Children With Allergic Rhinitis and Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, associate professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GuangzhouIRD-LSUN
Record Dates: First submitted 2015-01-21; First posted 2015-02-02 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Allergic Rhinitis; Inflammation; Respiratory Tract Diseases; Hypersensitivity
Keywords: allergic rhinitis；airway inflammation；hyperreactivity
MeSH Terms: conditions — Rhinitis, Allergic; Inflammation; Respiratory Tract Diseases; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide nasal spray (Active Comparator): Budesonide nasal spray ,64mcg/putt,1 spray/nostril, 2 times/day,for 12 consecutive weeks.
  Interventions: Drug: Budesonide nasal spray
- Placebo (Placebo Comparator): Placebo:nasal placebo spray,1spray/nostril, 2 times/day,for 12 consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide nasal spray — 64mcg/1putt, 1 putt/nostril,b.i.d
  Other Names: intanasal corticosteroids
  Arms: Budesonide nasal spray
Drug: Placebo — 1 putt/nostril,b.i.d
  Other Names: Placebo nasal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treating upper airway with intranasal corticosteroids in children with allergic rhinitis and no asthma may bring favors in reducing lower airway inflammation and improving small airway function.

DETAILED DESCRIPTION:
Type of study :

This is a prospective randomized,double-blind, placebo-controlled study , to clarity whether treating upper airway with intranasal corticosteroids in children with allergic rhinitis may bring favors in reducing elevated lower airway inflammation，improving airway reactivity and airway resistance.

Methods :

The children with allergic rhinitis accompanied lower airway inflammation such as elevated percentage of eosinophil in induced sputums and/or higher level of fractional exhaled nitric oxide(FeNO) are recruited.By using a random digit table, eligible subjects were randomized into one of two groups,to receive budesonide nasal spray (BUD group) or nasal placebo(placebo group), 1 spray/nostril, 2 times/day, for three consecutive months observation. The following measurements were performed: skin prick test (SPT), peripheral blood cells five-classification test, serum total immunoglobulin E (IgE) and specific IgE of common inhalant allergens testing, nasal lavage and inflammatory cells classification ，pulmonary function test, bronchial provocation test，airway resistance measured by impulse oscillation technique. Meanwhile,history of all subjects were collected, visual analogue scale，rhinitis symptoms scores and rhinoconjunctivitis quality of life questionnaire (RQLQ) scores were evaluated. Symptom scores and laboratory examinations are performed at baseline,4 w,8w and 12 w after treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of allergic rhinitis without asthma
* sensitized to more than 1 common aeroaller¬gens
* FeNO >20ppb and/or induced sputum Eosinophil>2.5%

Exclusion Criteria:

* Respiratory infection 2 weeks prior to initial visit
* children with nasal polyposis
* History of immunotherapy
* unable to complete the test or had limited understanding
* Use of systemic corticosteroids 4 weeks prior to initial visit
* nasal and inhaled corticosteroids 2 weeks prior to initial visit
* leukotriene receptor antagonists 2 weeks prior to initial visit
* Use of antihistamines 7 days prior to initial visit

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline fractional exhaled nitric oxide (FeNO) at 3 months | 3 months after treatment
  Fractional exhaled nitric oxide (FeNO) measured at 0 w,4 w,8 w and 12 w after treatment
Change from baseline eosinophils in sputum at 3 months | 3 months after treatment
  Eosinophils in sputum at measured at 0 w,4 w,8 w and 12 w after treatment

SECONDARY OUTCOMES:
Changes of lower airway resistance (Z5,R5,X5,R5-20,R20 and Fres) using impulse oscillation | 0 w,4 w,8 w and 12 w after treatment
Change of upper airway inflammation biomarker such as eosinophils in nasal lavage | 0 w,4 w,8 w and 12 w after treatment
Change of cumulative dosage of methacholine causing a 20% fall in forced expiratory volume in 1 second (PD20FEV1-MCH) | 0 w,4 w,8 w and 12 w after treatment
To measure the differences in nasal symptoms score (TSS) about groups after 12 weeks of therapy | 0 w,4 w,8 w and 12 w after treatment
  The parameters considered in the TSS were: nasal obstruction, sneezing, nasal discharge ,itching. These symptoms were scored: 0 = symptom absent, 1 = mild (symptoms present but not annoying), 2 = moderate (frequent and offensive symptoms but do not interfere with sleep or normal activities) 3 = severe (symptoms that interfere with sleep or normal activities).
The change in visual analogue scale score for symptoms of rhinitis | 0 w,4 w,8 w and 12 w after treatment
Juniper mini RQLQ | 0 w,4 w,8 w and 12 w after treatment
Change in levels of eosinophil（ECP），eosinophil peroxidase（EPO）, myeloperoxidase （MPO）and eosinophil-derived neurotoxin (EDN) in induced sputum and serum about groups after twelve weeks of therapy | At baseline and 12 w after treatment
Change in forced vital capacity (FVC) , in forced expiratory volume in 1 second (FEV1)，in forced expired flow at 25% of FVC(FEF25) and in forced expired flow at 75% of FVC (FEF75) about groups after twelve weeks of therapy. | 0 w,4 w,8 w and 12 w after treatment
Evaluation of the possible association between upper airway inflammation (eosinophil count in nasal lavage) and bronchial (PD20FEV1-MCH，FeNO and eosinophil count in induced sputum). | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Nanshanzhong Zhong, master, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China